CLINICAL TRIAL: NCT06865209
Title: Monolithic Zirconia Posterior Single Crowns. a Time-Efficiency Study of a Complete Digital Flow: a Randomized Clinical Trial.
Brief Title: Monolithic Zirconia Posterior Single Crowns: a Randomized Clinical Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Guillermo Galván Lobo, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 33/2020
Record Dates: First submitted 2021-01-24; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Posterior Single Edentulous Sites
Keywords: Single Posterior Implant Crowns; Cost Efficiency; Monolithic Zirconia Crowns; Full Digital Workflow; 3D Printed Prototype

STUDY DESIGN:
Intervention Model Description: Cost-efficiency study parallel study following CONSORT requisites
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, the care provider and the principal investigator will be masked through the entire process
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Finish Single Posterior Monolithic Zirconia Screw Retained Implant Crowns (Experimental): Direct finish single posterior monolithic zirconia screw retained implant crowns, performed with full digital flow direct finish prosthetic protocol.
  Interventions: Device: Monolithic Zirconia Posterior Single Screw Retained Implant Crowns
- 3d Prototype Guided Single Posterior Monolithic Zirconia Screw Retained Implant Crowns (Active Comparator): Direct finish single posterior monolithic zirconia screw retained implant crowns, performed with full digital flow direct finish prosthetic protocol.
  Interventions: Device: Monolithic Zirconia Posterior Single Screw Retained Implant Crowns

INTERVENTIONS:
Device: Monolithic Zirconia Posterior Single Screw Retained Implant Crowns — Posterior single edentulous sites will be rehabilitated with monolithic zirconia single posterior implant crowns following two different full digital workflows

SUMMARY:
Monolithic Zirconia Posterior Single Crown cost-efficiency study. Objective and subjective analysis will be performed through FIPS and PROMs scales to evaluate treatment quality outcomes.

DETAILED DESCRIPTION:
Introduction Posterior implant single crowns have become the treatment of choice for single tooth replacement in the posterior sectors, due to its biological implications and minimally invasive approach since it requires no preparation of the adjacent tooth and enabling a more efficient hygiene for the patient than a bridge restoration. However, implant-based restorations require more time and economical resources from the patient and the dentist compared to traditional teeth-supported restorations.

Currently the main interest is set upon broadening the potential patient spectrum for this kind of therapies, which can only be achieved by significally reducing the clinical treatment time and technical production time while maintaining an acceptable profit ratio and good quality treatment outcome.

Objectives The main goal of this study is to determine whether monolithic screw retained posterior implant crowns (test) are more time-efficient than metal ceramic screw retained posterior implant. Moreover, as secondary objectives every screw retained crown will be submitted for Functional Implant Prosthodontic Score (FIPS) and Patient Related Outcome Measures (PROMs) evaluation. Hypothesis Monolithic screw-retained posterior single implant crowns performed through a full digital workflow are more time-efficient than conventional-digital workflow fabricated metal-porcelain screw-retained posterior single implant crowns.

Monolitihic single posterior screw-retained implant crowns achieve better quality outcomes than metal porcelain single posterior screw-retained implant crowns.

Material & Methods A total of 40 implants placed at Master de Integrada de Adultos will participate in a time- efficiency study that will compare monolithic screw-retained posterior implant crowns to metal ceramic screw-retained posterior implant crowns ( gold standard), moreover, every restoration will be submitted for Functional Implant Prosthetic Score (FIPS) and Patient Related Outcome Measures (PROMs)

ELIGIBILITY:
Inclusion Criteria:

* Restorable implants
* No signs or previous history of periimplantitis
* Natural antagonist teeth
* Natural adjacent teeth

Exclusion Criteria:

* Non restorable implants
* Signs or previous history of periimplantitis
* No natural antagonist teeth
* No natural adjacent teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Cost | From the first visit to definitive crown placement
  Analyze how many cost units (monetary unit) are needed to make monolithic zirconia single posterior implant supported crowns to assess economic profitability of theses crowns
Efficiency | From the first visit to definitive crown placement
  Analyze how much time are needed to make monolithic zirconia single posterior implant supported crowns to assess economic profitability of theses crowns

SECONDARY OUTCOMES:
Functional Implant Prosthetic Score (FIPS) | 1 week post-op to 1 year follow up
  Analyze treatment quality outcomes according to the Functional Implant Prosthetic Score. Score 0-10
Patient Related Outcome Measures (PROMs) | 1 week post-op to 1 year follow up
  Analyze how the patient perceives treatment outcomes according to the Patient Related Outcome Measures scale. Score 0-10
Accuracy | Prosthetic Baseline to Definitive Crown Placement
  Analyze castless full digital workflow accuracy, comparing the matching accuracy of the definitive crowns to the digital wax up for both groups. Both STL meshes will be analyzed with Shape Designer by 3 Shape to asses how does the physical prostheses match the virtual wax ups

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontolico de Bellvitge Universidad de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brånemark PI, Zarb G, Albrektsson T, editors. Chicago: : Quintessence Publishing; 1985. Tissue-integrated prostheses: Osseointegration in clinical dentistry
- [Background] Mayer TM, Hawley CE, Gunsolley JC, Feldman S. The single-tooth implant: a viable alternative for single-tooth replacement. J Periodontol. 2002 Jul;73(7):687-93. doi: 10.1902/jop.2002.73.7.687. PMID 12146526
- [Background] Levin L, Sadet P, Grossmann Y. A retrospective evaluation of 1,387 single-tooth implants: a 6-year follow-up. J Periodontol. 2006 Dec;77(12):2080-3. doi: 10.1902/jop.2006.060220. PMID 17209794
- [Background] Muftu A, Chapman RJ. Replacing posterior teeth with freestanding implants: four-year prosthodontic results of a prospective study. J Am Dent Assoc. 1998 Aug;129(8):1097-102. doi: 10.14219/jada.archive.1998.0384. PMID 9715010
- [Background] Schwartz-Arad D, Samet N, Samet N. Single tooth replacement of missing molars: a retrospective study of 78 implants. J Periodontol. 1999 Apr;70(4):449-54. doi: 10.1902/jop.1999.70.4.449. PMID 10328659
- [Background] Jung SW, Lee JK, Um HS, Chang BS. A retrospective study on survival rate of the most posterior single tooth implant. J Korean Acad Periodontol. 2008;38:611-620.
- [Background] Salvi GE, Bragger U. Mechanical and technical risks in implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:69-85. PMID 19885435
- [Background] De Boever AL, Keersmaekers K, Vanmaele G, Kerschbaum T, Theuniers G, De Boever JA. Prosthetic complications in fixed endosseous implant-borne reconstructions after an observations period of at least 40 months. J Oral Rehabil. 2006 Nov;33(11):833-9. doi: 10.1111/j.1365-2842.2006.01638.x. PMID 17002743
- [Background] Vigolo P, Givani A, Majzoub Z, Cordioli G. Cemented versus screw-retained implant-supported single-tooth crowns: a 4-year prospective clinical study. Int J Oral Maxillofac Implants. 2004 Mar-Apr;19(2):260-5. PMID 15101598
- [Background] Nedir R, Bischof M, Szmukler-Moncler S, Belser UC, Samson J. Prosthetic complications with dental implants: from an up-to-8-year experience in private practice. Int J Oral Maxillofac Implants. 2006 Nov-Dec;21(6):919-28. PMID 17190302
- [Background] Bragger U, Aeschlimann S, Burgin W, Hammerle CH, Lang NP. Biological and technical complications and failures with fixed partial dentures (FPD) on implants and teeth after four to five years of function. Clin Oral Implants Res. 2001 Feb;12(1):26-34. doi: 10.1034/j.1600-0501.2001.012001026.x. PMID 11168268
- [Background] Sethi A, Kaus T, Sochor P, Axmann-Krcmar D, Chanavaz M. Evolution of the concept of angulated abutments in implant dentistry: 14-year clinical data. Implant Dent. 2002;11(1):41-51. doi: 10.1097/00008505-200201000-00013. PMID 11915544
- [Background] Koutouzis T, Wennstrom JL. Bone level changes at axial- and non-axial-positioned implants supporting fixed partial dentures. A 5-year retrospective longitudinal study. Clin Oral Implants Res. 2007 Oct;18(5):585-90. doi: 10.1111/j.1600-0501.2007.01386.x. Epub 2007 Jun 30. PMID 17608740
- [Background] Tawil G, Aboujaoude N, Younan R. Influence of prosthetic parameters on the survival and complication rates of short implants. Int J Oral Maxillofac Implants. 2006 Mar-Apr;21(2):275-82. PMID 16634499
- [Background] Rokni S, Todescan R, Watson P, Pharoah M, Adegbembo AO, Deporter D. An assessment of crown-to-root ratios with short sintered porous-surfaced implants supporting prostheses in partially edentulous patients. Int J Oral Maxillofac Implants. 2005 Jan-Feb;20(1):69-76. PMID 15747676
- [Background] Blanes RJ, Bernard JP, Blanes ZM, Belser UC. A 10-year prospective study of ITI dental implants placed in the posterior region. II: Influence of the crown-to-implant ratio and different prosthetic treatment modalities on crestal bone loss. Clin Oral Implants Res. 2007 Dec;18(6):707-14. doi: 10.1111/j.1600-0501.2006.01307.x. Epub 2007 Aug 13. PMID 17697000
- [Background] Del Corso M, Aba G, Vazquez L, Dargaud J, Dohan Ehrenfest DM. Optical three-dimensional scanning acquisition of the position of osseointegrated implants: an in vitro study to determine method accuracy and operational feasibility. Clin Implant Dent Relat Res. 2009 Sep;11(3):214-21. doi: 10.1111/j.1708-8208.2008.00106.x. Epub 2008 Jul 23. PMID 18657149
- [Background] Patzelt SB, Vonau S, Stampf S, Att W. Assessing the feasibility and accuracy of digitizing edentulous jaws. J Am Dent Assoc. 2013 Aug;144(8):914-20. doi: 10.14219/jada.archive.2013.0209. PMID 23904578
- [Background] Papaspyridakos P, Chen CJ, Gallucci GO, Doukoudakis A, Weber HP, Chronopoulos V. Accuracy of implant impressions for partially and completely edentulous patients: a systematic review. Int J Oral Maxillofac Implants. 2014 Jul-Aug;29(4):836-45. doi: 10.11607/jomi.3625. PMID 25032763
- [Background] Jeong ID, Lee JJ, Jeon JH, Kim JH, Kim HY, Kim WC. Accuracy of complete-arch model using an intraoral video scanner: An in vitro study. J Prosthet Dent. 2016 Jun;115(6):755-9. doi: 10.1016/j.prosdent.2015.11.007. Epub 2016 Jan 13. PMID 26794703
- [Background] Aragon ML, Pontes LF, Bichara LM, Flores-Mir C, Normando D. Validity and reliability of intraoral scanners compared to conventional gypsum models measurements: a systematic review. Eur J Orthod. 2016 Aug;38(4):429-34. doi: 10.1093/ejo/cjw033. Epub 2016 Jun 7. PMID 27266879
- [Background] Burzynski JA, Firestone AR, Beck FM, Fields HW Jr, Deguchi T. Comparison of digital intraoral scanners and alginate impressions: Time and patient satisfaction. Am J Orthod Dentofacial Orthop. 2018 Apr;153(4):534-541. doi: 10.1016/j.ajodo.2017.08.017. PMID 29602345
- [Background] Joda T, Bragger U. Patient-centered outcomes comparing digital and conventional implant impression procedures: a randomized crossover trial. Clin Oral Implants Res. 2016 Dec;27(12):e185-e189. doi: 10.1111/clr.12600. Epub 2015 Apr 12. PMID 25864771
- [Background] Zarone F, Russo S, Sorrentino R. From porcelain-fused-to-metal to zirconia: clinical and experimental considerations. Dent Mater. 2011 Jan;27(1):83-96. doi: 10.1016/j.dental.2010.10.024. Epub 2010 Nov 21. PMID 21094996
- [Background] Walton TR. A 10-year longitudinal study of fixed prosthodontics: clinical characteristics and outcome of single-unit metal-ceramic crowns. Int J Prosthodont. 1999 Nov-Dec;12(6):519-26. PMID 10815605
- [Background] Lin WS, Ercoli C, Feng C, Morton D. The effect of core material, veneering porcelain, and fabrication technique on the biaxial flexural strength and weibull analysis of selected dental ceramics. J Prosthodont. 2012 Jul;21(5):353-62. doi: 10.1111/j.1532-849X.2012.00845.x. Epub 2012 Mar 29. PMID 22462639
- [Background] Wettstein F, Sailer I, Roos M, Hammerle CH. Clinical study of the internal gaps of zirconia and metal frameworks for fixed partial dentures. Eur J Oral Sci. 2008 Jun;116(3):272-9. doi: 10.1111/j.1600-0722.2008.00527.x. PMID 18471247
- [Background] Land CH. Porcelain dental art: no.II. Dent Cosmos. 1903;45:615620.
- [Background] McLean JW, Hughes TH. The reinforcement of dental porcelain with ceramic oxides. Br Dent J. 1965 Sep 21;119(6):251-67. No abstract available. PMID 5212704
- [Background] Al-Amleh B, Lyons K, Swain M. Clinical trials in zirconia: a systematic review. J Oral Rehabil. 2010 Aug;37(8):641-52. doi: 10.1111/j.1365-2842.2010.02094.x. Epub 2010 Apr 9. PMID 20406352
- [Background] Piconi C, Maccauro G. Zirconia as a ceramic biomaterial. Biomaterials. 1999 Jan;20(1):1-25. doi: 10.1016/s0142-9612(98)00010-6. PMID 9916767
- [Background] Malkondu Ö, Tinastepe N, Akan E, et al. An overview of monolithic zirconia in dentistry. Biotechnol Biotechnol Equip. 2016;30:644-652.
- [Background] Sailer I, Muhlemann S, Fehmer V, Hammerle CHF, Benic GI. Randomized controlled clinical trial of digital and conventional workflows for the fabrication of zirconia-ceramic fixed partial dentures. Part I: Time efficiency of complete-arch digital scans versus conventional impressions. J Prosthet Dent. 2019 Jan;121(1):69-75. doi: 10.1016/j.prosdent.2018.04.021. Epub 2018 Jul 14. PMID 30017152